CLINICAL TRIAL: NCT03025074
Title: Virology, Immunology and Mechanisms of Liver Disease in Patients With Hepatitis C and Other Liver Diseases
Brief Title: Blood Collection Biorepository for Liver Disease Research
Status: Recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Andrew Talal, Professor of Medicine, State University of New York at Buffalo
Other Study IDs: Biobank Blood
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Non-Alcoholic Steatohepatitis(NASH); Hepatitis C; Hepatitis B; Fibrosis; Cirrhosis; Fatty Liver; Obesity, Childhood; Bariatric Surgery Candidate
Keywords: Liver Disease; Obesity; Hepatitis; HIV; Hepatology
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hepatitis C; Hepatitis B; Fibrosis; Fatty Liver; Pediatric Obesity; Liver Diseases; Obesity; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Serum, Plasma, Buffy Coat, Liver tissue (Core Needle Biopsy)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of establishing a biorepository is to provide high quality specimens (serum, plasma, buffy coat and liver tissue) for future researchers who are studying the effects that fatty liver and viral diseases have on the liver.

DETAILED DESCRIPTION:
The Biorepository at the University at Buffalo has been established to collect biological samples from patients with various types of liver disease. The objectives of this biorepository are to stimulate collaboration between clinicians and researchers, to bolster training of junior investigators and to promote multidisciplinary integration to advance translational medicine and to improve the health of patients all over the country. The purpose of this biorepository is to support investigators and to provide them with high quality specimens to promote their efforts in new discoveries or perfecting treatment of patients with liver diseases caused by Non-Alcoholic Fatty Liver Disease (NAFLD), Non-Alcoholic Steatohepatitis (NASH), Hepatitis C Virus (HCV), Hepatitis B Virus (HBV), and Human Immunodeficiency Virus (HIV). The goal is to obtain samples that represent patients seen in the clinics of medical centers in Western NY and from some of the rarer diseases encountered in these clinics. The ultimate goal is to develop the biorepository as Western New York's resource for clinically annotated human samples that can be used to conduct research that could lead to significant advances in patient care.

ELIGIBILITY:
Inclusion Criteria:

* This protocol is to establish a biobank of blood samples from individuals with or without liver diseases including viral hepatitis, liver cancer, NASH, and negative control samples.
* Children and teenagers will be special populations considered in this protocol.

Exclusion Criteria:

* Vulnerable populations such as adults unable to consent, infants, pregnant women or prisoners will not be considered for this research study.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with NASH, NAFLD, Fibrosis, Cirrhosis, Hepatitis B or C, HIV or any form of Liver Disease.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-07; Primary Completion 2099-12 (Estimated); Study Completion 2099-12 (Estimated)

PRIMARY OUTCOMES:
Number of samples collected | 52 weeks
  Total number of samples collected

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Talal, MD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo General Medical Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The Biorepository was created to provide high quality specimens to future researchers to advance their clinical and translational research.

REFERENCES:
- [Background] Zeremski M, Sylvester C, Talal AH. Response to Commentary on Zeremski et al. (2016): Improvements in HCV-related Knowledge Among Substance Users on Opioid Agonist Therapy After an Educational Intervention. J Addict Med. 2016 Sep-Oct;10(5):364-5. doi: 10.1097/ADM.0000000000000240. No abstract available. PMID 27685683
- [Background] Juluru K, Talal AH, Yantiss RK, Spincemaille P, Weidman EK, Giambrone AE, Jalili S, Sourbron SP, Dyke JP. Diagnostic accuracy of intracellular uptake rates calculated using dynamic Gd-EOB-DTPA-enhanced MRI for hepatic fibrosis stage. J Magn Reson Imaging. 2017 Apr;45(4):1177-1185. doi: 10.1002/jmri.25431. Epub 2016 Aug 16. PMID 27527820
- [Background] Zeremski M, Dimova RB, Pillardy J, de Jong YP, Jacobson IM, Talal AH. Fibrosis Progression in Patients With Chronic Hepatitis C Virus Infection. J Infect Dis. 2016 Oct 15;214(8):1164-70. doi: 10.1093/infdis/jiw332. Epub 2016 Aug 2. PMID 27485356
- [Background] Ocque AJ, Hagler CE, Difrancesco R, Woolwine-Cunningham Y, Bednasz CJ, Morse GD, Talal AH. Development and validation of a UPLC-MS/MS method for the simultaneous determination of paritaprevir and ritonavir in rat liver. Bioanalysis. 2016 Jul;8(13):1353-63. doi: 10.4155/bio-2016-0040. Epub 2016 Jun 9. PMID 27277877
- [Background] Zeremski M, Zavala R, Dimova RB, Chen Y, Kritz S, Sylvester C, Brown LS Jr, Talal AH. Improvements in HCV-related Knowledge Among Substance Users on Opioid Agonist Therapy After an Educational Intervention. J Addict Med. 2016 Mar-Apr;10(2):104-9. doi: 10.1097/ADM.0000000000000196. PMID 26881485
- [Background] Bednasz CJ, Sawyer JR, Martinez A, Rose PG, Sithole SS, Hamilton HR, Kaufman FS, Venuto CS, Ma Q, Talal A, Morse GD. Recent advances in management of the HIV/HCV coinfected patient. Future Virol. 2015;10(8):981-997. doi: 10.2217/fvl.15.64. PMID 26877758
- [Background] Cloherty G, Talal A, Coller K, Steinhart C, Hackett J Jr, Dawson G, Rockstroh J, Feld J. Role of Serologic and Molecular Diagnostic Assays in Identification and Management of Hepatitis C Virus Infection. J Clin Microbiol. 2016 Feb;54(2):265-73. doi: 10.1128/JCM.02407-15. Epub 2015 Dec 9. PMID 26659219
- [Background] Zeremski M, Dimova RB, Benjamin S, Penney MS, Botfield MC, Talal AH. Intrahepatic and Peripheral CXCL10 Expression in Hepatitis C Virus-Infected Patients Treated With Telaprevir, Pegylated Interferon, and Ribavirin. J Infect Dis. 2015 Jun 1;211(11):1795-9. doi: 10.1093/infdis/jiu807. Epub 2014 Dec 15. PMID 25512630